CLINICAL TRIAL: NCT00949377
Title: Can Methylnaltrexone Safely Treat Opioid Related Constipation in the Emergency Department?
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit enough patients at a single center.
Sponsor: Beth Israel Medical Center (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 064-09
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-04

CONDITIONS: Colonic Inertia
Keywords: Constipation; opioid
MeSH Terms: conditions — Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylnaltrexone Bromide (Experimental)
  Interventions: Drug: Methylnaltrexone Bromide (MNTX)
- Normal Saline (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylnaltrexone Bromide (MNTX) — The recommended dose of MNTX (Relistor) is 8 mg for patients weighing 38 kg to less than 62 kg (84 lbs to less than 136 lbs) or 12 mg for patients weighing 62 kg to 114 kg (136 lbs to 251 lbs). Patients whose weight is below 38 kg or greater than 114 kg, will be dosed at 0.15 mg/kg.
  Other Names: Relistor
  Arms: Methylnaltrexone Bromide
Drug: Placebo — Normal saline
  Arms: Normal Saline

SUMMARY:
The investigators want to prove that people WITHOUT advanced cancer who are taking opioid medications (for problems like back pain) can receive methylnaltrexone (MNTX) safely. Since the FDA has only approved MNTX for advanced cancer patients, the investigators' research is investigating how MNTX can work for NON-cancer patients. This research is being conducted to prove that MNTX can work for non-cancer patients with opioid related constipation.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 and greater
2. Clinical diagnosis of constipation
3. Any patients that report taking an opioid analgesic for greater than two (2) weeks (eg known oncology patients and chronic pain syndrome patients, including those with low back pain or sciatica)
4. Patients must have previously tried a stable laxative regiment for at least three (3) days prior to study entry.
5. All patients will have a flat and upright abdominal x-ray, and chest x-ray to exclude gastrointestinal (GI) obstruction. Any patients who have radiographic evidence of GI obstruction will need a CT scan of the abdomen to exclude GI obstruction prior to study enrollment.
6. Females of childbearing potential must have a negative pregnancy test and must be encouraged to use appropriate birth control for a period after the study.
7. Willing to comply with study instructions and sign an informed consent

Exclusion Criteria:

1. Pregnancy or lactation
2. Recent surgery within six (6) weeks of the emergency department visit
3. Opioid withdrawal syndrome as determined by clinical judgment.
4. Patients with previous history of diabetic gastroparesis.
5. Any patient who has known or suspected gastrointestinal obstruction
6. Any patients with creatinine clearance ≤ 30 mL/min
7. Constipation for which other medical causes cannot be excluded such as anticholinergic medications, botulinum toxin, or botulism.
8. Any patient with SBP ≤ 80 mmHg or DBP ≤ 45 mmHg or unstable vital signs.
9. Inability to understand or follow the instructions associated with the clinical study as determined by clinical judgment.
10. A known history of substance abuse on methadone maintenance therapy > 12 months
11. Allergy or contraindication to use of methylnaltrexone
12. Prior enrollment in study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Laxation | 4 hours

SECONDARY OUTCOMES:
Opioid withdrawal symptoms | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Lemeneh Tefera, MD, Principal Investigator — Beth Israel Medical Center; Michael Heller, MD, Study Director — Beth Israel Medical Center